CLINICAL TRIAL: NCT06250621
Title: Manual or Digitally Guided Surgical Technique for Replacing Single Tooth Edentulism by Means of Sub-crestally Placed Implants. A 3-year Parallel Randomized Clinical Study on Marginal Bone Levels Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Santi Paolo e Carlo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC 1564/18
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: Dental Implant; Marginal Bone Loss; Peri Implant Health; Supral Tissue Height

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (GD) (Experimental): in this group were considered implant sites treated with a digitally guided surgery procedure
  Interventions: Procedure: Implant placement
- Control Group (FH) (Active Comparator): in this group were considered implant sites treated without a digitally guided surgery procedure
  Interventions: Procedure: Implant placement

INTERVENTIONS:
Procedure: Implant placement — Implants were placed by means of a template for a guided surgery approach (GD Group) or with a standard free-hand surgical approach without any additional device (FH Group). A non expert doctor (less that 20 implants placed in the professional activity) was selected for the procedures related to the GD Group; a skilled operator (more than 1000 implants placed in the professional activity) was selected for the procedures related to the FH Group, respectively.
  A two-stage surgical technique was chosen. Implants were placed (Anyridge, Megagen Implants, Seoul, Korea) 1 mm below the crestal level, as recommended by the manufacturer. After flap elevation the height of the supra-crestal soft tissue (STH) was measured by means of a calibrated probe.
  An inter-implant distance of 3 mm at least, and/or an interproximal space from 1.5 to 3 mm between an implant and the adjacent tooth were observed.
  Flaps were sutured over the implants to allow a submerged healing.

SUMMARY:
The aim of the present prospective study was to investigate after a 2-year of follow-up any influence of the surgical technique, manual or digitally guided, on peri-implant marginal bone levels stability in implants placed 1 mm sub-crestally.

Patients were treated by means of platform-switched implants provided with a 5 degrees internal conical connection and supporting single screw-retained fixed crowns. Marginal bone level (MBL) measured at prosthesis installation (t0) at 1 (t1), 2 (t2) and at 3 years of follow-up visit (t3) were considered. MBL change from t0 to t3 was investigated. The distance between the implant neck and the first radiographically detected bone to implant contact was considered to evaluate the bone loss. Two groups were considered: Test Group (GD) for implant sites treated with a digitally guided surgery procedure. Control Group (FH) for implants surgically placed without digitally guided surgery, respectively. All the procedures were performed by an experienced operator. Additionally, for both groups MBL changes were correlated to different supra-crestal soft tissue height (STH) amounts: less than 3 and ≥ 3 millimeters, respectively. Peri-implant soft tissue parameters such as probing depth (PPD), modified Sulcus Bleeding Index (mBI) and modified Plaque Index (mPI), were assessed for all the restorations included.

ELIGIBILITY:
Inclusion Criteria:

* absence of mandibular and/or maxillary atrophy; presence of partial edentulism of at least one pair of elements and adequate amount of bone tissue to be able to insert an implant, i.e., a minimum amount of residual bone of 5 mm in thickness and 10 mm in height; presence of an antagonistic element with respect to the tooth to be rehabilitated.

Exclusion Criteria:

* patients presenting with a clinical history of systemic diseases and metabolic deficits, presence or previous leukocyte dysfunction/deficiency, blood disorders, hemophilia, dicoumarolic drug therapy, treatment of prolonged steroid therapy, history of neoplasms resulting in chemotherapy and/or radiation therapy in the head and neck district, history of chronic renal problems, chronic liver disease, bone metabolism disorders, uncontrolled endocrine disorders, and ongoing pregnancy and/or lactation. presence of local inflammation such as untreated periodontitis, bruxism condition or clenching habit, habitual oral infections, mucosal disorders (erosive lichen planus), oral lesions (ulcers, malignant lesions), inadequate oral hygiene, and poor compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Marginal bone loss | From t0 to t3 (3-years of follow up)
  Measurements were made at mesial and distal aspect of each implant and were reported in millimeters.
  Because of implants were sub-crestally positioned, measurements where bone was under the implant to abutment level were classified as negative values. On the contrary, measurements where implant neck was over the bone crest were classified as positive values.
  Measurements were made at mesial and distal aspect of each implant and were reported in millimeters.
  Because of implants were sub-crestally positioned, measurements where bone was under the implant to abutment level were classified as negative values. On the contrary, measurements where implant neck was over the bone crest were classified as positive values.

SECONDARY OUTCOMES:
STH | During surgery
  After flap elevation the height of the supra-crestal soft tissue (STH) was measured by means of a calibrated probe.

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio ER Romeo, Prof., Study Director — Odontostomatologia I, ASST Santi Paolo e Carlo, P.O. S. Paolo
Locations (1):
- ASST Santi Paolo e Carlo, Milan, MI, Italy